CLINICAL TRIAL: NCT00274105
Title: A Double Blind, 2:1 Randomised Monocentre Study to Investigate the Efficacy and Safety of Telmisartan (80 mg qd) Concerning the Amelioration of Structural Alterations and Function of Endothelium in Cardiovascular Risk Patients (SAFE-CRP: Structural Alterations and Function of Endothelium in Cardiovascular Risk Patients)
Brief Title: SAFE-CRP: Structural Alterations and Function of Endothelium in Cardiovascular Risk Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.350
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Coronary Arteriosclerosis
MeSH Terms: conditions — Hypertension; Coronary Artery Disease | interventions — Telmisartan

INTERVENTIONS:
Drug: telmisartan
Drug: Placebo

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of telmisartan 80 mg administered once daily in patients with documented coronary artery disease (CAD) and a probably cardiovascular risk profile concerning the amelioration of structural alterations and endothelial function.

The primary objective of this trial is to evaluate the efficacy in particular with regard to the percentage change of atheroma volume in the femoral artery.The secondary objective is to evaluate the change in the plaque size- assessed by intravascular ultrasound, the increase in Flow Dependent Dilation provoked by intraarterial infusion of three increasing concentrations of Acetylcholine, and the change in seated systolic blood pressure.

Endothelial dysfunction is a primary event in atherogenesis and all known cardiovascular risk factors have been associated with endothelial dysfunction before atherosclerotic vascular disease manifests itself clinically. Pivotal to endothelial dysfunction is a disturbance in the function of endothelium-derived nitric oxide (NO). Recently, it could be shown that acute and chronic angiotensin-1 receptor antagonism reversed endothelial dysfunction in atherosclerosis. In experimental atherosclerosis, AT1 receptor blockade appears to have protective effects. Respective potential mechanisms include the prevention of endothelial injury, the augmentation of NO activity, the inhibition of lipid peroxidation and an antiproliferative effect. These findings together with the most recent data that losartan improves endothelial function and NO activity suggest that AT1 receptor antagonism may also be antiatherogenic in patients with atherosclerosis. Angiotensin II influences smooth muscle cell migration, hyperplasia, and hypertrophy. Angiotensin II also enhances production of local superoxide anion, which will inactivate nitric oxide. Inhibition of these reactions by the AT1-Blocker telmisartan may therefore interfere with atherosclerotic plaque formation.

DETAILED DESCRIPTION:
Methodology:

2:1 randomised, double-blind and placebo-controlled parallel-group design

Planned/actual number of subjects:

Enrolled: 30/33, randomised: 30/22, completed: 30/15

Duration of treatment:

9 months: telmisartan (80 mg) or Placebo (80 mg)

Study Hypothesis:

The trial is designed as a group comparison of telmisartan 80 mg and placebo, where the treatment groups are randomised in 2:1 relation, to investigate the efficacy of telmisartan on structural alterations and endothelial dysfunction as measured as the percentage change from baseline after 36 weeks of treatment of the atheroma volume in the femoral artery using IVUS .

Secondary endpoints are the changes from baseline in the flow dependent dilatation after a acetylcholine challenge which follows a nitro-glycerin bolus, the change of the total atheroma volume, the percentage atheroma volume measured by intravascular ultrasound (IVUS) and the infalmmatory parameters MCP-1, CRP, ox LDL antibodies and sPLA2 activity and amount.

In an analysis of covariance using baseline as covariate all endpoints will be investigated. If the assumptions of normal distribution are not fulfilled, nonparametric methods will be applied (Wilcoxon-Mann-Whitney test).

Comparison(s):

Placebo 80 mg

ELIGIBILITY:
Inclusion criteria:

1. > 35 years of age
2. History of coronary artery disease (CAD)
3. Ability to provide written informed consent

Exclusion criteria:

1. Pre-menopausal women (last menstruation < 1 year prior to start of the screening visit) who:

   1. are not surgically sterile; and/or
   2. are nursing
   3. are of child-bearing potential and are NOT practising acceptable means of birth control, do NOT plan to continue using this method throughout the study and do NOT agree to submit to periodic pregnancy testing during participation in studies of > 3-months duration. Acceptable methods of birth control include oral, implantable or injectable contraceptives
2. Diastolic blood pressure > 110 mmHg or systolic blood pressure > 180 mmHg at any visit during the study (run-in or randomised period)
3. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   1. SGPT(ALT) or SGOT(AST) > than 2 times the upper limit of normal range
   2. Serum creatinine > 2.3 mg/dL
4. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, patients post-renal transplant or with only one kidney
5. Clinically relevant hypokalaemia or hyperkalaemia
6. Uncorrected volume depletion
7. Uncorrected sodium depletion
8. Primary aldosteronism
9. Hereditary fructose intolerance
10. Biliary obstructive disorders
11. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists
12. History of drug or alcohol dependency within 6 months
13. Chronic administration of any medications known to affect blood pressure, except medication allowed by the protocol
14. Any investigational therapy within one month of signing the informed consent form
15. Known hypersensitivity to any component of the formulation
16. Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of telmisartan
17. Stroke within the last 6 months
18. Myocardial infarction within the last 30 days
19. Cardiac surgery within the last 3 months
20. Hyperthyroidosis
21. Hemodynamically relevant valvular disease
22. Restrictive hypertrophic cardiomyopathy
23. Unstable angina pectoris
24. CAD with the indication of bypass surgery.

Min Age: 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2001-03-01 (Actual); Primary Completion 2004-10-01 (Actual); Study Completion 2004-10-01 (Actual)

PRIMARY OUTCOMES:
Change of intima/media ratio in the femoral artery measured by intravascular ultrasound (IVUS) | after 39 weeks

SECONDARY OUTCOMES:
Change in plaque size in the femoral artery measured by IVUS | after 39 weeks
Increase in FDD (Flow dependent dilation) stimulated by intra-arterial infusion of Acetylcholine (ACH) | after 39 weeks
Change in serum inflammatory markers (CRP, MCP-1, oxLDL antibodies, and VCAM) | after 39 weeks
Change in seated blood pressure (BP) at trough | after 39 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (2):
- Germany (2):
  - Universitätsklinikum Charité, Berlin
  - Med. Hochschule Hannover, Hanover

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency